CLINICAL TRIAL: NCT02237196
Title: Anti-TSLP (AMG 157) Plus Antigen-Specific Immunotherapy for Induction of Tolerance in Individuals With Cat Allergy (ITN057AD)
Brief Title: Anti-TSLP (AMG 157) Plus Antigen-Specific Immunotherapy for Induction of Tolerance in Individuals With Cat Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN057AD; CATNIP (Other: Immune Tolerance Network)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Cat Allergy; Cat Hypersensitivity
Keywords: cat-allergic; cat immunotherapy; anti-thymic stromal lymphopoietin (anti-TSLP)
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AMG 157+Cat Immunotherapy (Experimental): AMG 157 will be administered every four weeks.
  Cat immunotherapy will be administered weekly.
  Interventions: Biological: AMG 157; Biological: Cat Immunotherapy
- AMG 157 Placebo+Cat Immunotherapy (Active Comparator): Placebo for AMG 157 of similar appearance will be administered every four weeks.
  Cat immunotherapy will be administered weekly.
  Interventions: Biological: Cat Immunotherapy; Biological: AMG 157 Placebo
- AMG 157+Cat Immunotherapy Placebo (Experimental): AMG 157 will be administered every four weeks.
  Placebo for Cat immunotherapy will be administered weekly.
  Interventions: Biological: AMG 157; Biological: Cat Immunotherapy Placebo
- Placebo-Placebo (Placebo Comparator): Placebo for AMG 157 will be administered every four weeks.
  Placebo for cat immunotherapy will be administered weekly.
  Interventions: Biological: Cat Immunotherapy Placebo; Biological: AMG 157 Placebo

INTERVENTIONS:
Biological: AMG 157 — AMG 157 will be administered once every 4 weeks at dose of 700 mg intravenously. Each AMG 157 dose will be administered at least 1 day before immunotherapy through week 24, then on the same day as immunotherapy thereafter.
  Other Names: MEDI9929/AMG 157
  Arms: AMG 157+Cat Immunotherapy; AMG 157+Cat Immunotherapy Placebo
Biological: Cat Immunotherapy — A standardized allergen extract licensed in the United States for allergen immunotherapy, and is formulated as a long-acting suspension for subcutaneous injection
  Other Names: Cat Allergen Extract
  Arms: AMG 157 Placebo+Cat Immunotherapy; AMG 157+Cat Immunotherapy
Biological: Cat Immunotherapy Placebo — Placebo for allergen-specific immunotherapy administered subcutaneously
  Other Names: Placebo for Cat Immunotherapy
  Arms: AMG 157+Cat Immunotherapy Placebo; Placebo-Placebo
Biological: AMG 157 Placebo — Placebo for AMG 157 administered intravenously
  Other Names: Placebo for AMG157
  Arms: AMG 157 Placebo+Cat Immunotherapy; Placebo-Placebo

SUMMARY:
This trial will test whether a novel therapeutic approach, cat immunotherapy combined with an investigational new drug called MEDI9929/AMG 157 (an anti-TSLP [thymic stromal lymphopoietin] antibody being co-developed by Amgen and MedImmune) can lead to lasting tolerance to cat allergen.The objective of the study is to determine whether one year of immunotherapy combined with MEDI9929/AMG 157 can induce tolerance to cat allergen.

DETAILED DESCRIPTION:
This study will implement the concept referred to as "allergen-plus," which aims to enhance the disease-modifying mechanisms of allergen-specific immunotherapy by combining it with other anti-inflammatory or immune-modulating agents. Thymic stromal lymphopoietin (TSLP) is a cytokine which appears to be instrumental in both initiating and maintaining allergic sensitivity to antigens, and Immune Tolerance Network (ITN) investigators hypothesize that blocking TSLP during the administration of cat immunotherapy will induce durable immune changes that lead to tolerance.

CATNIP will be conducted at multiple sites in the US and enroll cat-allergic adults who will be randomized to four possible treatment groups: immunotherapy plus MEDI9929/AMG 157, immunotherapy plus placebo, placebo plus MEDI9929/AMG 157, or two corresponding placebos. This study is specifically enrolling cat allergic individuals who do not live with cats in order to limit exposure to the allergen outside of the study. Treatment will be given for about one year, followed by one year off therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate-severe allergic rhinitis caused by cat exposure for at least 2 yrs
* Skin prick test wheal >/=5 mm to standardized cat extract
* Immunoglobulin E (IgE) >/=0.7 kU/L (class 2) to cat extract
* Screening nasal allergen challenge in which:

  *TNSS is </= 3 after the 0 concentration (vehicle control only) dose,
* TNSS increase is </=1 from the TNSS prior to allergen administration to the TNSS after the 0 concentration (vehicle control only) dose,

  * TNSS is >/=8 after the highest dose, and
  * Between the first non-zero dose and 10 minutes after the highest dose,either:
* >/=3 sneezes are counted or
* >20% drop in PNIF is recorded
* Body mass index (BMI) between 1 and 32 kg/m^2, inclusive at screening
* Clinically acceptable physical examination and electrocardiogram (ECG) results (12-lead reporting RR, PR, QRS, QT and QTcF) prior to Day 0 based on the opinion of the investigator
* Adequate renal function (defined by creatinine clearance >80 mL/min using the Cockcroft Gault equation)
* For women of childbearing age, a willingness to use a highly effective form of contraception for five months after last dose of study medication. Highly effective methods of birth control include abstinence, vasectomy by the male partner, or a condom with spermicide in combination with either hormonal birth control, IUD or barrier methods used by the woman.
* For men with female partners of childbearing potential, agreement not to donate sperm and to inform their female partner of their participation in this clinical study and use highly effective methods of birth control for five months after last dose of study medication. Highly effective methods of birth control include abstinence, vasectomy, or a condom with spermicide in combination with either hormonal birth control, Intrauterine device (IUD) or barrier methods used by the woman.
* The ability to give informed consent and comply with study procedures

Exclusion Criteria:

* Prebronchodilator Forced Expiratory Volume at one second (FEV1) less than 0% of predicted value at screening visit
* History of moderate or higher Allergic Rhinitis and its Impact on Asthma (ARIA) severity classification for allergic rhinitis in the last year due to allergens other than cat
* History of asthma meeting the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report 3 (EPR3) classification of mild-persistent or worse in the past year, other than with cat exposure, requiring regular inhaled corticosteroids for >4 weeks per year
* History of serious chronic medical conditions which might interfere with treatment or assessments
* History of emergency visit or hospital admission for asthma in the previous 12 months
* History of chronic obstructive pulmonary disease (COPD)
* History of significant recurrent acute sinusitis, defined as 2 episodes/yr for the last 2 years, all of which required antibiotic treatment
* History of chronic sinusitis, defined as a sinus symptoms lasting >12 weeks that includes >/=2 major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, purulent or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, and ear pain, pressure, or fullness.
* History of systemic disease affecting the immune system such as autoimmune diseases, immune complex disease, or immunodeficiency, where, in the opinion of the study physician, participation in the trial would pose a risk or significant effect on the immune system
* Diabetes (Type I or II)
* Evidence of any active or suspected bacterial, viral, fungal or parasitic infection(s) within 30 days prior to randomization
* High risk of parasitic disease as judged by the investigator
* Positive QuantiFERON(R) tuberculin test UNLESS the potential subject has been treated with appropriate chemoprophylaxis
* Exposure to an individual with active tuberculosis within six months from randomization
* Subjects tested positive for HIV antibody, Hep B surface antigen, or Hep C antibody
* At randomization, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
* History of malignancy of any type, including basal cell and squamous cell cancers of the skin, within 5 years of enrollment
* Tobacco smoking (ANY) within the last year or a history of >/=10 pack years
* Previous immunotherapy treatment with cat allergen within the previous 10 yrs
* Any history of grade 4 anaphylaxis due to any cause as defined by the CTCAE grading criteria for immunotherapy
* History of bleeding disorders or treatment with anticoagulation therapy
* Treatment with omalizumab within 6 months prior to randomization
* Currently taking any of the following medications: beta blockers; tricyclic antidepressants; monoamine oxidase inhibitors; or anti-IgE monoclonal antibody treatment
* Ongoing systemic immunosuppressive treatment
* History of intolerance to the study therapy, rescue medications, or their excipients
* For women of childbearing age a positive serum or urine pregnancy test with sensitivity of <50 mIU/mL within 72 hours before the start of study therapy
* The use of any investigational drug within 6 months of randomization
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Corren, MD, Study Chair — University of California, Los Angeles
Locations (9):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Asthma & Allergy Center, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - ASTHMA Inc. Clinical Research Center, Seattle, Washington
  - University Wisconsin, Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in upon completion of the study in: 1.)ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.)TrialShare, a clinical trials research portal developed by the Immune Tolerance Network that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Derived] Corren J, Larson D, Altman MC, Segnitz RM, Avila PC, Greenberger PA, Baroody F, Moss MH, Nelson H, Burbank AJ, Hernandez ML, Peden D, Saini S, Tilles S, Hussain I, Whitehouse D, Qin T, Villarreal M, Sever M, Wheatley LM, Nepom GT, Sanda S; Immune Tolerance Network ITN057AD CATNIP Study Team. Effects of combination treatment with tezepelumab and allergen immunotherapy on nasal responses to allergen: A randomized controlled trial. J Allergy Clin Immunol. 2023 Jan;151(1):192-201. doi: 10.1016/j.jaci.2022.08.029. Epub 2022 Oct 9. PMID 36223848
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) Website — http://www.immunetolerance.org/
- See also: World Allergy Organization (WAO) Subcutaneous Immunotherapy Systemic Reaction Grading System — https://www.aaaai.org/practice-resources/practice-tools/immunotherapy-forms/immunotherapy-systemic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ages 18 years to 65 years with a history of moderate to severe allergic rhinitis caused by cat exposure were recruited from 9 clinical centers in the United States from March 3, 2015 to March 21, 2017.
Groups:
- AMG 157+Cat Immunotherapy: AMG 157 will be administered every four weeks.
  Cat immunotherapy will be administered weekly.
  AMG 157: AMG 157 will be administered once every 4 weeks at dose of 700 mg intravenously. Each AMG 157 dose will be administered at least 1 day before immunotherapy through week 24, then on the same day as immunotherapy thereafter.
  Cat Immunotherapy: A standardized allergen extract licensed in the United States for allergen immunotherapy, and is formulated as a long-acting suspension for subcutaneous injection
- AMG 157 Placebo+Cat Immunotherapy: Placebo for AMG 157 of similar appearance will be administered every four weeks.
  Cat immunotherapy will be administered weekly.
  Cat Immunotherapy: A standardized allergen extract licensed in the United States for allergen immunotherapy, and is formulated as a long-acting suspension for subcutaneous injection
  AMG 157 Placebo: Placebo for AMG 157 administered intravenously
- AMG 157+Cat Immunotherapy Placebo: AMG 157 will be administered every four weeks.
  Placebo for Cat immunotherapy will be administered weekly.
  AMG 157: AMG 157 will be administered once every 4 weeks at dose of 700 mg intravenously. Each AMG 157 dose will be administered at least 1 day before immunotherapy through week 24, then on the same day as immunotherapy thereafter.
  Cat Immunotherapy Placebo: Placebo for allergen-specific immunotherapy administered subcutaneously
- Placebo-Placebo: Placebo for AMG 157 will be administered every four weeks.
  Placebo for cat immunotherapy will be administered weekly.
  Cat Immunotherapy Placebo: Placebo for allergen-specific immunotherapy administered subcutaneously
  AMG 157 Placebo: Placebo for AMG 157 administered intravenously
Period: Overall Study
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Started | 32 | 31 | 30 | 28
Completed | 24 | 25 | 20 | 17
Not Completed | 8 | 6 | 10 | 11
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 4 | 2 | 4 | 6
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 1
Not completed — Site Error | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo | Total
Number analyzed (Participants) | 32 | 31 | 30 | 28 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 1 | 5
  Between 18 and 65 years | 30 | 29 | 30 | 27 | 116
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.52) | 30.4 (8.86) | 31.9 (9.92) | 30.5 (10.91) | 30.5 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 16 | 15 | 75
  Male | 8 | 11 | 14 | 13 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 5 | 15
  Not Hispanic or Latino | 29 | 27 | 27 | 22 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 1 | 3 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 0 | 7
  White | 21 | 28 | 24 | 24 | 97
  More than one race | 2 | 0 | 0 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 31 | 30 | 28 | 121

OUTCOME MEASURES:

1. Primary Outcome: Total Nasal Symptom Score (TNSS) Area Under the Curve (AUC)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring nasal congestion and blockade, rhinorrhea, itching, and sneezing. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Higher scores indicate more severe nasal symptoms. The trapezoidal rule was used to calculate the TNSS AUC. The primary outcome compared the mean TNSS AUC from 0 to 1 hour after cat Nasal Allergen Challenge at 104 weeks by treatment group, using a longitudinal repeated measures model in the ITT sample. The model included fixed effects for treatment, time, and treatment by time interaction and included covariates for site, baseline TNSS AUC and Baseline Cat exposure (low vs high). The primary endpoint was assessed at week 104 using a contrast in least squares means between the following groups: AMG 157+Cat Immunotherapy and AMG 157 Placebo+Cat Immunotherapy.
Time Frame: 0 to 1 hour of the NAC at Week 104
Population: Intent-to-treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Total Nasal Symptom Score * Hour
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
Total Nasal Symptom Score * Hour | 2.46 [1.73 to 3.19] | 2.81 [2.13 to 3.49] | 3.66 [2.74 to 4.59] | 3.10 [2.11 to 4.10]
Statistical Analysis 1: Comparison: AMG 157+Cat Immunotherapy vs AMG 157 Placebo+Cat Immunotherapy; Test type: Superiority; p = 0.314, Longitudinal repeated measures analysis; Model adjusts for Site, Baseline TNSS AUC, and Baseline Cat exposure (low vs high); Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.51 to 0.49], Standard Error of Mean 0.5038

2. Secondary Outcome: Skin Prick Test Endpoint Titration
Description: A dilution series of standardized cat allergen extracts were applied in duplicate on the participant's upper back. Wheal size was assessed 15 minutes after application.
Time Frame: 15 minutes after Time 0 of the skin prick titration test at: Baseline (Week 0) and Weeks 1, 4, 12, 26, 52, 78 and 104
Population: A cross-sectional analysis of the observed measures within the intent-to-treat population was used in the reporting of secondary endpoints.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
mm
  Baseline | 45.11 [40.74 to 49.49] | 46.29 [38.88 to 53.69] | 45.01 [40.17 to 49.84] | 44.49 [38.25 to 50.73]
  Week 1: number analyzed (Participants) | 29 | 27 | 27 | 26
  Week 1 | 45.92 [38.08 to 53.77] | 50.25 [42.22 to 58.28] | 43.33 [38.20 to 48.47] | 44.06 [38.31 to 49.82]
  Week 4: number analyzed (Participants) | 28 | 26 | 27 | 27
  Week 4 | 39.24 [33.48 to 45.00] | 35.44 [29.39 to 41.49] | 44.01 [38.56 to 49.47] | 41.58 [35.59 to 47.57]
  Week 12: number analyzed (Participants) | 29 | 24 | 24 | 23
  Week 12 | 30.12 [23.94 to 36.30] | 22.08 [16.33 to 27.84] | 45.85 [40.13 to 51.57] | 44.74 [39.09 to 50.38]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | 21.96 [16.41 to 27.51] | 22.21 [14.45 to 29.98] | 43.93 [38.13 to 49.72] | 43.40 [37.27 to 49.53]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 21.34 [15.48 to 27.19] | 16.84 [12.69 to 20.99] | 34.92 [27.39 to 42.45] | 39.64 [30.51 to 48.77]
  Week 78: number analyzed (Participants) | 25 | 25 | 22 | 18
  Week 78 | 22.21 [16.31 to 28.11] | 25.13 [20.18 to 30.08] | 32.28 [24.67 to 39.90] | 39.32 [30.39 to 48.25]
  Week 104: number analyzed (Participants) | 24 | 25 | 19 | 17
  Week 104 | 26.88 [19.95 to 33.81] | 26.67 [21.68 to 31.66] | 39.82 [32.24 to 47.39] | 36.19 [29.33 to 43.06]

3. Secondary Outcome: Skin Early Phase Response (EPR) to Intradermal Testing
Description: Concentrations of standardized cat hair extract were applied intradermally to the forearm. Wheal size was measured 15 minutes and 6 hours after application. The Early Phase Response (EPR) is the response measured at 15 minutes after application.
Time Frame: 15 minutes after Time 0 of the intradermal test at: Baseline (Week 0) and Weeks 26, 52, and 104
Population: A cross-sectional analysis of the observed measures within the intent-to-treat was used in the reporting of secondary endpoints.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
mm
  Baseline | 16.05 [15.25 to 16.8] | 15.34 [14.42 to 16.26] | 15.98 [15.12 to 16.85] | 16.52 [15.66 to 17.37]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | 11.21 [10.13 to 12.29] | 11.65 [10.86 to 12.43] | 14.15 [13.09 to 15.21] | 14.64 [13.21 to 16.07]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 10.65 [9.53 to 11.78] | 10.69 [9.72 to 11.67] | 13.35 [12.33 to 14.36] | 14.21 [12.40 to 16.03]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | 11.04 [9.80 to 12.28] | 12.09 [10.80 to 13.38] | 12.63 [11.55 to 13.70] | 13.21 [11.60 to 14.82]

4. Secondary Outcome: Skin Late Phase Response (LPR) to Intradermal Testing
Description: Concentrations of standardized cat hair extract were applied intradermally to the forearm. Wheal size was measured 15 minutes and 6 hours after application. The Late Phase Response (LPR) is the response measured at 6 hours after application.
Time Frame: 6 hours status post cat allergen challenge at: Baseline (Time 0) and Weeks 26, 52 and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 29 | 28 | 27 | 27
mm
  Baseline | 32.62 [26.62 to 38.62] | 23.41 [17.23 to 29.59] | 27.22 [19.33 to 35.11] | 34.65 [27.27 to 42.03]
  Week 26: number analyzed (Participants) | 27 | 27 | 27 | 25
  Week 26 | 13.50 [8.41 to 18.59] | 13.83 [8.93 to 18.74] | 26.44 [18.68 to 34.20] | 31.28 [23.01 to 39.55]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 13.67 [9.17 to 18.18] | 10.06 [6.12 to 13.99] | 23.23 [16.17 to 30.28] | 29.36 [18.62 to 40.10]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | 15.58 [11.05 to 20.12] | 14.48 [10.37 to 18.59] | 25.40 [18.27 to 32.53] | 32.38 [21.08 to 43.68]

5. Secondary Outcome: Peak Total Nasal Symptom Score (TNSS): Early Phase Response (EPR)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring nasal congestion and blockade, rhinorrhea, itching, and sneezing. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Higher scores indicate more severe nasal symptoms. Peak TNSS EPR is the highest value recorded between 0 and 1 hour inclusive.
Time Frame: 0 to 1 hour of the NAC at: Baseline (Week 0) and Weeks 26, 52, 78 and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Peak Total Nasal Symptom Score
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
Peak Total Nasal Symptom Score
  Baseline | 9.31 [8.92 to 9.71] | 9.52 [9.05 to 9.98] | 9.17 [8.76 to 9.57] | 8.96 [8.59 to 9.34]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | 3.64 [2.74 to 4.55] | 5.41 [4.30 to 6.52] | 6.78 [5.63 to 7.92] | 7.96 [7.04 to 8.88]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 3.04 [2.16 to 3.91] | 4.73 [3.63 to 5.83] | 6.09 [4.78 to 7.39] | 6.75 [5.72 to 7.78]
  Week 78: number analyzed (Participants) | 25 | 25 | 22 | 18
  Week 78 | 4.24 [3.33 to 5.15] | 4.80 [3.63 to 5.97] | 6.82 [5.32 to 8.32] | 5.83 [4.58 to 7.09]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | 4.67 [3.59 to 5.74] | 6.16 [5.13 to 7.19] | 6.85 [5.30 to 8.40] | 6.12 [4.46 to 7.77]

6. Secondary Outcome: Total Nasal Symptom Score (TNSS) Early Phase Response (EPR)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring nasal congestion and blockade, rhinorrhea, itching, and sneezing. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Higher scores indicate more severe nasal symptoms. The trapezoidal rule was used to calculate the TNSS AUC. The Early Phase Response (EPR) is the TNSS AUC from 0 to 1 hour.
Time Frame: 0 to 1 hour of the NAC at: Baseline (Week 0) and Weeks 26, 52, 78 and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Total Nasal Symptom Score * Hour
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
Total Nasal Symptom Score * Hour
  Baseline | 5.49 [4.99 to 6.00] | 5.59 [5.00 to 6.18] | 4.91 [4.27 to 5.55] | 5.55 [4.96 to 6.15]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | 1.83 [1.36 to 2.29] | 2.71 [2.13 to 3.30] | 3.38 [2.69 to 4.08] | 4.09 [3.44 to 4.74]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 1.53 [1.03 to 2.03] | 2.34 [1.74 to 2.93] | 3.07 [2.33 to 3.81] | 3.77 [2.99 to 4.55]
  Week 78: number analyzed (Participants) | 25 | 25 | 22 | 18
  Week 78 | 2.04 [1.42 to 2.66] | 2.31 [1.45 to 3.17] | 3.23 [2.37 to 4.09] | 2.88 [1.93 to 3.84]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | 2.46 [1.73 to 3.19] | 2.81 [2.13 to 3.49] | 3.66 [2.74 to 4.59] | 3.10 [2.11 to 4.10]

7. Secondary Outcome: Total Nasal Symptom Score (TNSS) Late Phase Response (LPR)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring nasal congestion and blockade, rhinorrhea, itching, and sneezing. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Higher scores indicate more severe nasal symptoms. The trapezoidal rule was used to calculate the TNSS AUC. The Late Phase Response (LPR) is the TNSS AUC from 5 to 6 hours.
Time Frame: Hours 5 to 6 of the NAC at: Baseline (Week 0) and Weeks 26, 52, and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Total Nasal Symptom Score * Hour
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
Total Nasal Symptom Score * Hour
  Baseline | 1.36 [0.86 to 1.86] | 1.52 [0.86 to 2.17] | 1.13 [0.70 to 1.57] | 1.25 [0.81 to 1.69]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | 0.30 [0.13 to 0.47] | 0.67 [0.29 to 1.05] | 0.54 [0.11 to 0.97] | 0.90 [0.50 to 1.30]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | 0.48 [0.18 to 0.78] | 0.60 [0.20 to 0.99] | 0.24 [0.06 to 0.42] | 0.73 [0.14 to 1.31]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | 0.69 [0.21 to 1.17] | 1.02 [0.26 to 1.78] | 0.53 [0.20 to 0.85] | 0.76 [-0.17 to 1.70]

8. Secondary Outcome: Peak Nasal Inspiratory Flow (PNIF) Early Phase Response (EPR) Area Under the Curve (AUC)
Description: PNIF is defined as the speed of inspiration of air in Liters per minute when breathing in into the lungs through the nose. Lower scores indicate less ability to breathe air into the lungs due to more severe nasal symptoms. The Early Phase Response (EPR) is the PNIF AUC from 0 to 1 hour of the NAC.
Time Frame: 0 to 1 hour of the NAC at: Baseline (Week 0) and Weeks 26, 52 and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: L/min * Hour
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
L/min * Hour
  Baseline | -15.14 [-25.62 to -4.66] | -10.66 [-20.28 to -1.04] | -12.48 [-24.05 to -0.91] | -10.25 [-20.01 to -0.49]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | -2.88 [-11.19 to 5.44] | 2.26 [-6.53 to 11.05] | -11.04 [-20.13 to -1.95] | -8.02 [-22.30 to 6.26]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | -8.65 [-19.69 to 2.39] | -4.90 [-14.67 to 4.86] | -0.80 [-10.86 to 9.25] | -8.70 [-17.90 to 0.50]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | -11.35 [-25.34 to 2.63] | -11.90 [-23.05 to -0.75] | -9.13 [-24.08 to 5.83] | -13.09 [-30.47 to 4.30]

9. Secondary Outcome: Peak Nasal Inspiratory Flow (PNIF) Late Phase Response (LPR) Area Under Curve AUC
Description: PNIF is defined as the speed of inspiration of air in Liters per minute when breathing in into the lungs through the nose. Lower scores indicate less ability to breathe air into the lungs due to more severe nasal symptoms. The Late Phase Response (LPR) is the PNIF AUC from hours 5 to 6 of the NAC.
Time Frame: Hours 5 to 6 of the NAC at: Baseline (Week 0) and Weeks 26, 52, 78, and 104
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: L/min * Hour
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
Number analyzed (Participants) | 32 | 31 | 30 | 28
L/min * Hour
  Baseline | -52.24 [-64.31 to -40.17] | -53.44 [-63.87 to 43.00] | -42.49 [-53.30 to -31.68] | -50.03 [-62.32 to -37.74]
  Week 26: number analyzed (Participants) | 28 | 27 | 27 | 25
  Week 26 | -18.34 [-29.10 to -7.57] | -17.35 [-26.53 to -8.17] | -40.42 [-52.09 to -28.75] | -53.97 [-68.85 to -39.09]
  Week 52: number analyzed (Participants) | 26 | 26 | 23 | 20
  Week 52 | -25.29 [-38.24 to 12.35] | -23.42 [-33.78 to -13.07] | -35.87 [-51.51 to -20.24] | -44.71 [-54.89 to -34.53]
  Week 78: number analyzed (Participants) | 25 | 25 | 22 | 18
  Week 78 | -31.93 [-42.14 to 21.73] | -24.55 [-36.66 to 12.44] | -37.56 [-52.55 to -22.57] | -42.26 [-59.70 to -24.81]
  Week 104: number analyzed (Participants) | 24 | 25 | 20 | 17
  Week 104 | -43.41 [-61.54 to -25.29] | -35.98 [-49.21 to -22.75] | -49.01 [-62.18 to -35.84] | -52.42 [-69.07 to -35.77]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Total number at risk is reported for the Safety population;one participant was randomized and discontinued prior to starting Study Therapy,thus not included in the Safety population.
  1. Local reactions/AEs:FDA Guidance,Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (Sep 2007) 2. Systemic AEs:WAO Subcutaneous Immunotherapy Systemic Reaction Grading System 3.Other AE's: NCI Common Terminology Criteria for Adverse Events (V4.03).
Groups:
- AMG 157+Cat Immunotherapy: AMG 157 administered every four weeks and Cat immunotherapy administered weekly
- AMG 157 Placebo+Cat Immunotherapy: Placebo for AMG 157 administered every four weeks and Cat immunotherapy administered weekly
- AMG 157+Cat Immunotherapy Placebo: AMG 157 administered every four weeks and Placebo for Cat immunotherapy administered weekly
- Placebo-Placebo: Placebo for AMG 157 administered every four weeks and Placebo for Cat immunotherapy administered weekly
Arm/Group | AMG 157+Cat Immunotherapy | AMG 157 Placebo+Cat Immunotherapy | AMG 157+Cat Immunotherapy Placebo | Placebo-Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/32 | 3/31 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 25/32 | 18/31 | 18/29 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG 157+Cat Immunotherapy (N=32) | AMG 157 Placebo+Cat Immunotherapy (N=31) | AMG 157+Cat Immunotherapy Placebo (N=29) | Placebo-Placebo (N=28)
All-Cause Mortality (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG 157+Cat Immunotherapy (N=32) | AMG 157 Placebo+Cat Immunotherapy (N=31) | AMG 157+Cat Immunotherapy Placebo (N=29) | Placebo-Placebo (N=28)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypersensitivity (Immune system disorders) | 6 (36) | 3 (8) | 1 (1) | 1 (2)
Injection site hypersensitivity (Immune system disorders) | 8 (12) | 3 (4) | 2 (2) | 1 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (14) | 4 (7) | 9 (17) | 9 (16)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 6 (9) | 5 (10) | 6 (7)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (7) | 0 (0) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (12) | 2 (15) | 3 (4)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
None listed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT02237196/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02237196/SAP_001.pdf